CLINICAL TRIAL: NCT06693453
Title: Evaluating the Effects of Electronic Acupuncture Combined With Dry Cupping Therapy in Treating Back Pain Due to Lumbar Spondylosis in the qi Stagnation and Blood Stasis Pattern: A Randomized Clinical Trial
Brief Title: Effects of Electronic Acupuncture Combined With Dry Cupping Therapy in Treating Back Pain Due to Lumbar Spondylosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, NGUYEN THI THUY AN, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1099/HDDD-DHYD
Record Dates: First submitted 2024-11-06; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Back Pain
Keywords: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Group (Sham Comparator): Sham Coparator: 38 patients were treated with acupuncture using Khanh Phong 20x15 needles inserted into specific acupuncture points. Afterward, the acupuncture needles were connected to electrodes to administer electrical stimulation through the KWD808-1 electroacupuncture machine. The Sham group will receive placebo dry cupping therapy using two size 1 acrylic cups (internal diameter 4.5 cm), with a distance of 3 cm between each cup, placed parallel to the spine, bilaterally along the boundaries of acupoints BL17, BL23, and B25. This group will undergo placebo dry cupping therapy for 7 minutes, every 4 days (3 sessions over 2 weeks). However, the cups will be prepared with small holes <2 mm in diameter to release the negative pressure within seconds. Double-sided tape will be used to ensure the cups remain attached and in contact with the skin.
  Interventions: Other: Electroacupuncture and Sham Dry cupping
- Intervention Group (Experimental): 38 patients were treated with acupuncture using Khanh Phong 20x15 needles inserted into specific acupuncture points. Afterward, the acupuncture needles were connected to electrodes to administer electrical stimulation through the KWD808-1 electroacupuncture machine. Dry cupping will be applied using 6 size 1 acrylic cups (internal diameter 4.5 cm), with a distance of 3 cm between each cup, parallel to the spine, bilaterally according to the boundaries of acupoints BL17, BL23, and B25. This group will perform electroacupuncture for 20 minutes daily (10 sessions over 2 weeks) and dry cupping for 10 minutes every 4 days (3 sessions over 2 weeks).
  Interventions: Other: Electroacupuncture and Dry cupping

INTERVENTIONS:
Other: Electroacupuncture and Dry cupping — This group will perform electroacupuncture for 20 minutes daily (10 sessions over 2 weeks) and dry cupping for 7 minutes every 4 days (3 sessions over 2 weeks)
  Arms: Intervention Group
Other: Electroacupuncture and Sham Dry cupping — This group will perform Electroacupuncture for 20 minutes daily (10 sessions over 2 weeks) and Sham Dry cupping for 7 minutes every 4 days (3 sessions over 2 weeks)
  Arms: Sham Group

SUMMARY:
The goal of this clinical trial is to learn if Electroacupuncture combined with Dry cupping therapy works to treat back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern. I

The main questions it aims to answer are:

* Does Electroacupuncture combined with Dry cupping therapy reduces pain on Visual Analog Scale (VAS) of patients suffered from back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern?
* Dose Electroacupuncture combined with Dry cupping therapy improving the daily activities on Oswestry Disability index (ODI) of patients suffered from back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern?
* What medical problems do participants have when taking Electroacupuncture combined with Dry cupping therapy ? Researchers will compare dry cupping to a sham dry cupping (a sham cupping device was developed by establishing a small hole to reduce the negative pressure after suction such that inner pressure could not be maintained in the cup) to see if dry cupping therapy works to treat back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern.

Patients with back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern will be registered for this study. They will be treated with a combination of Electroacupuncture combined with Dry cupping therapy.

The intervention period is two weeks. Electronic acupuncture will be performed once a day for 2 weeks. Dry cupping therapy will be performed every 4 days for 2 weeks. Data on the Visual Analog Scale (VAS), Oswestry Disability index (ODI), and side effects of Electroacupuncture and Dry cuppingwill be recorded before the study and weekly for 2 weeks.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if Electroacupuncture combined with Dry cupping therapy works to treat back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern. I

The main questions it aims to answer are:

* Does Electroacupuncture combined with Dry cupping therapy reduces pain on Visual Analog Scale (VAS) of patients suffered from back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern?
* Dose Electroacupuncture combined with Dry cupping therapy improving the daily activities on Oswestry Disability index (ODI) of patients suffered from back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern?
* What medical problems do participants have when taking Electroacupuncture combined with Dry cupping therapy ? Researchers will compare dry cupping to a sham dry cupping (a sham cupping device was developed by establishing a small hole to reduce the negative pressure after suction such that inner pressure could not be maintained in the cup) to see if dry cupping therapy works to treat back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern.

Patients with back pain due to lumbar spondylosis in the qi stagnation and blood stasis pattern will be registered for this study. They will be treated with a combination of Electroacupuncture combined with Dry cupping therapy.

The intervention period is two weeks. Electronic acupuncture will be performed once a day for 2 weeks. Dry cupping therapy will be performed every 4 days for 2 weeks. Data on the Visual Analog Scale (VAS), Oswestry Disability index (ODI), and side effects of Electroacupuncture and Dry cuppingwill be recorded before the study and weekly for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, male and female, 18-70 years of age.
* Report pain intensity between 3 and 7 according to the pain numerical rating scale.
* ODI disability index ≥10%.
* Patients diagnosed with lower back pain due to Qi stagnation and blood stasis syndrome (diagnosed by a Traditional Medicine Doctor) with clinical signs: stabbing, fixed lower back pain, worse at night, stiffness in the lumbar region, difficulty bending forward, extending, or rotating. The tongue is dark purple, possibly with blood stasis spots, and the pulse is wiry and tight or hesitant.

Exclusion Criteria:

* Have previously performed cupping therapy in some body segment;
* Present neurological, vestibular, visual or auditory deficits that make assessments impossible;
* Being in the gestational period;
* Having severe spinal disease (including fractures, tumour, inflammatory diseases, or tumours);
* Have undergone previous spinal surgery;
* Present with radiating or sacroiliac back pain; another rheumatic disease such as fibromyalgia,or ankylosing spondylitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Disability - ODI | baseline and week 2
  The Oswestry Disability Index (ODI) questionnaire will be used to analyze disability in people with low back pain.This instrument contains 10 items that assess the impact of low back pain on various functional activities. Values range from 0 to 5, with the highest value indicating greater disability. The final result is the sum of all items. The validated version in Portuguese is used.

SECONDARY OUTCOMES:
Change in Visual Analog Scale (VAS) | baseline and week 2
  Pain will be measured using the Visual Analog Scale (VAS). Patients will be asked to circle a number from 0 to 10, where 0 represents "no pain" and 10 represents "the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ho Chi Minh University of Medicine and Phamacy, Ho Chi Minh City,, Ho Chi Minh City, Vietnam